CLINICAL TRIAL: NCT06913413
Title: Effects Of 8-Week Core Stabilization Exercise With Vitamin D On Pain and Functional Limitation in Adults With Chronic Non-Specific Low Back Pain
Brief Title: Effects Of 8-Week Core Stabilization Exercise With Vitamin D On Pain and Functional Limitation in Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MSRSW/Batch-Fall23/796
Record Dates: First submitted 2025-03-29; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- core stabilization exercise (Experimental)
  Interventions: Combination Product: core stabilization exercise
- stabilization exercise (Active Comparator)
  Interventions: Diagnostic Test: stabilization exercise

INTERVENTIONS:
Combination Product: core stabilization exercise — Will receive 8 week core stabilization exercise 3 session per week which include 10 min warm up and 10 min cool down (walking ) 6 sets of movements co contraction of abdominal muscles (Abdominal hollowing) ,bridging ,dead bug ,plank with 50,000 IU of vitamin D weekly
  Arms: core stabilization exercise
Diagnostic Test: stabilization exercise — stabilization exercise 3 session per week which include 10 min warm and 10 min cool down (walking ) sham medicine, 6 sets of movements co contraction of abdominal muscles (Abdominal hollowing) ,bridging ,dead bug and plank
  Arms: stabilization exercise

SUMMARY:
Chronic non-specific low back pain (CNSLBP) is a prevalent condition contributing to pain, functional limitations, and reduced quality of life. Core stabilization exercises (CSE) have shown promise in enhancing spinal stability and reducing symptoms. Additionally, vitamin D supplementation plays a critical role in musculoskeletal health. Study objective will be to determine combined effect of vitamin D supplementation and core Stabilization exercises is better than core Stabilization Exercises alone in reducing pain-related and functional independence among chronic non-specific low back patient A randomized controlled trial will be conducted on 52 adults aged 25-45 diagnosed with Chronic non-specific low back pain.

DETAILED DESCRIPTION:
Subjects will be divided into two groups: the intervention group will receive an 8-week Core stabilization exercises program alongside daily vitamin D supplementation, while the control group will receive either Core stabilization exercises alone Visual Analog Scale (VAS), and Oswestry Disability

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 25 to 45 years will be included.
* Both gender Male /Female will participate.
* Subjects with diagnosed non-specific low lumber pain persisting for at least 12 weeks will be included.
* Subjects must have baseline pain score of ≥4 on the Visual Analog Scale.
* Confirmed serum vitamin D levels <30 ng/m will be included

Exclusion Criteria:

* Low lumber pain due to specific causes such as fracture malignancy infection or inflammatory diseases (e.g. ankylosing spondylitis).
* Presence of significant comorbidities that could interfere with participation (e.g. cardiovascular neurological or respiratory disorders).
* History of spinal surgery within the last year.
* Subjects currently taking vitamin D supplements or undergoing other treatments for vitamin D deficiency.
* Use of medications such as corticosteroids or opioids that might affect pain perception or functional assessment.
* Enrolled in any other physical therapy or pain management program within the last three months.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
The Visual Analogue Scale (VAS) | 12 Months
  The Visual Analogue Scale (VAS) uses a 10 cm line with anchors like "no pain" and "worst pain imaginable", and the score is determined by measuring the distance (in mm or cm) from the "no pain" end to the patient's mark, ranging from 0 to 100
The Oswestry Disability Index (ODI) | 12 Months
  The Oswestry Disability Index (ODI) is a questionnaire used to assess functional disability in individuals with low back pain, with scores ranging from 0% (no disability) to 100% (maximum disability), and interpreted as follows: 0-20% minimal disability, 21-40% moderate, 41-60% severe, 61-80% crippling, and 81-100% bed-bound or exaggerated symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Shoukat Hospital Near Session Court Jhang Road Chiniot, Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No